CLINICAL TRIAL: NCT07403305
Title: The Effect of Water Physical Exercise Program in Thermal Water and Hydropinotherapy on Cardiovascular Health
Acronym: WPEPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Bragança (Other)
Collaborators: Universidade do Porto (Other); Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Anna Carolina Cortez Ribeiro, Principal Investigator, Instituto Politécnico de Bragança
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPBraganca; UIDB/00690/2020; UIDP/00690 (Other Grant/Funding Number: Fundação para Ciência e Tecnologia); LA/P/0007/2020 (Other Grant/Funding Number: Fundação para Ciência e Tecnologia); UIDB/00617/2020, LA/P/0064/202 (Other Grant/Funding Number: Fundação para Ciência e Tecnologia (FCT)); PRT/BD/154584/2023 (Other Grant/Funding Number: Fundação para Ciência e Tecnologia (FCT))
Record Dates: First submitted 2026-01-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular (CV) Risk
Keywords: Thermal Water; Water Exercise; Hydropinotherapy; Lipid Profile; Cardiovascular Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I: Control (No Intervention): Control
- Arm II: WPEP in thermal water (Other): Water Physical Exercise Program in thermal water
  Interventions: Behavioral: WPEP in thermal water
- Arm III: Hydropinotherapy (Other): Hydropinotherapy with thermal water combined with bay leaf (L. nobilis)
  Interventions: Other: Hydropinotherapy
- Arm IV: WPEP in thermal water + Hydropinotherapy (Other): Water Physical Exercise Program in thermal water in thermal water and hydropinotherapy with thermal water combined with bay leaf (L. nobilis)
  Interventions: Behavioral: WPEP in thermal water; Other: Hydropinotherapy

INTERVENTIONS:
Behavioral: WPEP in thermal water — Water Physical Exercise Program (WPEP) in thermal water The classes will take place in water maintained at 34°C. Training sessions will occur twice a week, with 50 minutes each and classes limited to 20 participants. Dumbbells and flotation devices will be used to increase exercise resistance, focusing on three main areas: upper body, lower body, and cardiorespiratory and abdominal exercises.
  Each session will begin with a 5-10-minute active warm-up period. The main workout will consist of a high-intensity interval training protocol with multi-joint exercises. The session will conclude with a 5-10-minute cool-down period. All sessions will be supervised and led by experienced exercise physiologists and physiotherapists to ensure participant safety and exercise efficacy.
  Arms: Arm II: WPEP in thermal water; Arm IV: WPEP in thermal water + Hydropinotherapy
Other: Hydropinotherapy — The hydropinotherapy intervention consists of the oral ingestion of thermal water combined with bay leaf (Laurus nobilis). Participants assigned to this intervention will ingest 200 mL of Chaves thermal water infused with dried bay leaf (L. nobilis) twice per week. The infusion will be prepared by the research team by adding 5 g of dried bay leaf (L. nobilis) to the thermal water and allowing it to infuse for 15 minutes, followed by filtration through a strainer. All participants will be observed by the research team during ingestion to ensure compliance and safety.
  The thermal water used in this intervention is natural mineral water from Termas de Chaves, which emerges at a temperature of 77.0°C. It is classified as gasocarbonic, sodium bicarbonate, fluoride-based, and highly mineralized, with bicarbonate, chloride, sodium, and potassium as the predominant ions.
  Arms: Arm III: Hydropinotherapy; Arm IV: WPEP in thermal water + Hydropinotherapy

SUMMARY:
The goal of this randomized four-arm clinical trial is to determine the effect of 16-week water physical exercise program in thermal water and hydroponotherapy on lipide profile in middle-aged and elderly people, with controlled health conditions.

Participants will be randomizate into four arms:

* Arm I: Control
* Arm II: Water Physical Exercise Program (WPEP) in thermal water
* Arm III: Hydropinotherapy with thermal water combined with bay leaf (L. nobilis)
* Arm IV: WPEP in thermal water and hydropinotherapy with thermal water combined with bay leaf (L. nobilis)

Primary outcome:

1. Lipid profile (cholesterol total, low-density lipoprotein cholesterol (c-LDL), high-density lipoprotein cholesterol (c-HDL), triglycerides)

   Secondary parameters:
2. Inflammatory biomarkers: interleukin-6 (IL-6), C-reactive protein (CRP)
3. Glucose metabolisc: fasting plasma glucose, insulin, Hemoglobin A1c (HbA1c)
4. Aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, bilirubin, creatinine.
5. Anthropometric and clinical variables: weight, waist to hip ratio, body composition and bone mineral density
6. Systolic and diastolic blood pressure
7. Physical function
8. Lifestyle parameters: sleep quality, quality of life and eating habits

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age: >45 years
* Written informed consent prior to participation
* Physical condition suitable for participating in physical exercise activities
* Controlled health conditions

Exclusion Criteria:

* History of chronic or severe diseases that may affect study outcomes or limit study participation, such as:
* Decompensated cardiovascular disease, renal insufficiency, or severe liver disease
* Conditions preventing the ability in physical activity (e.g., severe respiratory issues, reduced mobility, severe arthritis)
* Severe psychiatric or cognitive disorders that could affect comprehension or adherence to the study
* Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) or corticosteroids
* Pregnancy or lactation
* Less than 80% attendance at the 16-week aquatic exercise program

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Lipid profile (total cholesterol, HDL-C, LDL-C, triglycerides) | 16 weeks
  Change in total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and triglyceride concentrations (mg/dL), measured by enzymatic spectrophotometry, with LDL-C calculated.

SECONDARY OUTCOMES:
Interleukin-6 (IL-6) | 16 weeks
  Change in serum interleukin-6 (IL-6) concentration (pg/mL), measured by enzyme-linked immunosorbent assay (ELISA)
C-reactive protein (CRP) | 16 weeks
  Change in serum C-reactive protein concentration (mg/L) measured by chemiluminescent microparticle immunoassay (CMIA).
Plasma Glucose | 16 weeks
  Change in fasting plasma glucose concentration (mg/dL), measured using standard laboratory methods.
Insulin | 16 weeks
  Change in fasting serum insulin concentration (µIU/mL), measured using standard laboratory methods.
Hemoglobin A1C (HbA1c) | 16 weeks
  Change in glycated hemoglobin (HbA1c, %), measured using standard laboratory methods.
Hepatic enzymes | 16 weeks
  Change in serum aspartate transaminase (AST) activity (U/L), alanine transaminase (ALT) activity (U/L), measured by enzymatic spectrophotometry.
Bilirubin | 16 weeks
  Change in total bilirubin concentration (mg/dL), measured by enzymatic spectrophotometry.
Blood pressure | 16 weeks
  Change in systolic and diastolic blood pressure (mmHg), measured using a digital blood pressure monitor following a standardized seated protocol, with the average of two readings recorded.
Waist and hip circumferences | 16 weeks
  Change in waist circumference (cm) and hip circumference (cm), measured using a non-elastic measuring tape according to ISAK protocols.
Body composition | 16 weeks
  Change in total fat mass (kg), truncal fat mass (kg), abdominal fat mass (kg), lean body mass (kg), assessed by dual-energy X-ray absorptiometry (DXA).
Bone mineral density | 16 weeks
  Change in bone mineral density (g/cm²) from baseline to 16 weeks, assessed by dual-energy X-ray absorptiometry (DXA).
Maximal oxygen uptake (VO₂ max) | 16 weeks
  Change in maximal oxygen uptake (mL/kg/min), assessed using a graded treadmill exercise test to volitional exhaustion.
Isokinetic muscle strength | 16 weeks
  Change in peak torque (Nm) of knee flexors and extensors, hip flexors/extensors and abductors/adductors, and ankle dorsiflexors and plantarflexors, assessed using isokinetic dynamometry.
Sleep quality | 16 weeks
  Change in sleep quality score, assessed by the Pittsburgh Sleep Quality Index (PSQI; score range 0-21, higher scores indicate worse sleep quality).
Health-related quality of life | 16 weeks
  Change in health-related quality of life score from baseline to 16 weeks, assessed by the Short Form-36 Health Survey (SF-36; score range 0-100, higher scores indicate better health status).
Pain intensity | 16 weeks
  Change in pain intensity score from baseline to 16 weeks, assessed by the Numeric Rating Scale (NRS; score range 0-10, higher scores indicate worse pain).
Psychosocial risk factors | 16 weeks
  Change in psychosocial risk classification from baseline to 16 weeks, assessed by the Start Back Screening Tool (SBST; score range 0-9, higher scores indicate higher psychosocial risk).
Total energy intake | 16 weeks
  Change in total energy intake (kcal/day), assessed using a 24-hour dietary recall administered by a trained nutritionist.
Macronutrient intake | 16 weeks
  Change in macronutrient intake (g/day: proteins, total fats, carbohydrates, fiber), assessed using a 24-hour dietary recall administered by a trained nutritionist.

IPD SHARING:
Plan to Share IPD: No